CLINICAL TRIAL: NCT00108420
Title: Prazosin Treatment for Combat Trauma PTSD Nightmares and Sleep Disturbance
Brief Title: Prazosin Treatment for Combat Trauma PTSD (Post-Traumatic Stress Disorder) Nightmares and Sleep Disturbance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-018-02F
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Stress Disorder, Post-Traumatic
Keywords: Prazosin; Stress Disorders, Post-traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Prazosin

INTERVENTIONS:
Drug: Prazosin

SUMMARY:
The purpose of this study is to determine whether prazosin will reduce the incidence of nightmares, sleep disturbance, and overall symptoms in combat trauma-exposed individuals with PTSD.

DETAILED DESCRIPTION:
The combat stress-related nightmares and sleep disturbance that often follow exposure to military combat are distressing and frequently persistent symptoms that impair quality of life and both occupational and social (e.g., family) function. One of the most frequently reported and most troubling symptoms of PTSD is trauma-content nightmares. These nighttime symptoms have been notoriously resistant to treatment with psychotropic medications such as anxiolytics, the SSRIs, and sedating antihistamines such as cyproheptadine. The SSRIs sertraline (Zoloft®) and paroxetine (Paxil®) are the only drugs FDA approved for PTSD. This approval was based on modest overall PTSD improvement compared to placebo in large multicenter trials that enrolled almost exclusively noncombat trauma subjects. Placebo-controlled SSRI trials for PTSD in combat veterans have been negative or equivocal.

Neurobiologic data suggest that combat stress-related nightmares and sleep disturbance in PTSD are related to enhanced central nervous system (CNS) adrenergic activity, particularly at night. Prazosin is a CNS-active, non-sedating alpha-1 antagonist that has long been generically available for the treatment of hypertension and benign prostatic hypertrophy. We recently demonstrated in Vietnam combat veterans with chronic PTSD that prazosin is robustly effective for previously treatment refractory combat trauma related nightmares, sleep disturbance and overall PTSD severity and functional impairment.

The goal of this study is to evaluate the efficacy and tolerability of prazosin compared to placebo for combat stress-related nightmares, sleep disturbance and overall function in combat-trauma exposed persons with PTSD.

Primary outcome measures will be Clinical Global Impression of Change, Recurrent Distressing Dreams and Difficulty Falling and Staying Asleep items of the CAPS, total CAPS (exclusive of the dreams and sleep items), and the Pittsburgh Sleep Quality Index. Depression and quality of life also will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Combat-trauma exposed persons with a diagnosis of PTSD
* No diagnosis of lifetime schizophrenia, schizoaffective disorder, bipolar disorder, psychotic disorder, or any DSM-IV cognitive disorder; current delirium, or substance dependence disorder within 3 months of the study or current substance use other than alcohol (no more than 2 drinks/day); severe psychiatric instability or situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to patient or others
* In good general medical health (no acute or significant chronic medical illness, including unstable angina, recent myocardial infarction, history of congestive heart failure, preexisting hypotension [systolic <110] or orthostatic hypotension [systolic drop > 20 mmHg after two minutes standing or any drop with dizziness]; insulin-dependent diabetes mellitus; chronic renal or hepatic failure, pancreatitis, gout, Meniere's disease, benign positional vertigo, narcolepsy, allergy or previous adverse reaction to prazosin or other alpha-1 antagonist, or any unstable medical condition).
* Stable dose of nonexcluded medications for concurrent stable medical conditions for at least 4 weeks prior to randomization.
* Specific criteria used to validate presence of combat stress-related nightmares and sleep disturbance will include: score > 5 (of a maximum score of 8) on the CAPS Recurrent Distressing Dreams item. (CAPS score >5 places subjects in the upper third of nightmare severity) or score > 5 (of a maximum score of 8) on the CAPS Difficulty Falling or Staying Asleep item.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Study Completion 2007-03

PRIMARY OUTCOMES:
Clinical Global Impression of Change
Recurrent Distressing Dreams and Difficulty Falling and Staying Asleep items of the CAPS
Total CAPS (exclusive of the dreams and sleep items)
The Pittsburgh Sleep Quality Index
Depression
Quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States